CLINICAL TRIAL: NCT02422862
Title: Clinical Effects of Upper Cervical Translatoric Mobilization in Patients With Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Miguel Malo Urriés, PhD, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMU.01.001
Record Dates: First submitted 2015-04-13; First posted 2015-04-21 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Headache
Keywords: Physiotherapy; Manual Therapy
MeSH Terms: conditions — Headache

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- UC-TSM (Experimental): Upper cervical translatoric spinal mobilization (UC-TSM). UC-TSM is a physical therapy technique used to improve range of movement, consisting on a manual stretching of the cervical spine of the patient during 30 minutes.
  Interventions: Other: UC-TSM
- Control (No Intervention): The control group receive no treatment intervention during 30 minutes (a similar time as the UC-TSM group).

INTERVENTIONS:
Other: UC-TSM — Upper cervical translatoric spinal mobilization: a 30 minutes treatment consisting of 30" series of translatoric mobilizations of the upper cervical spine with 10" rest between sets. For that purpose, the patient is positioned in supine, with the cervical spine in neutral position. The therapist place a hand dorsally at the level of the vertebral arch of C1 with the metacarpophalangeal and radial border of the index finger. The other hand is placed posteriorly under the occiput, with the shoulder positioned anteriorly on the patient's forehead. The mobilization force is directed dorsally from the shoulder until the therapist feel a marked resistance and then apply slightly more pressure in order to perform a stretching mobilization.
  Arms: UC-TSM

SUMMARY:
Frequently, headache is associated with disorders of the cervical spine, specially on the upper cervical spine. Therefore, restoration of the upper cervical mobility is considered fundamental for the treatment of headache.

Manual therapy interventions seek to restore upper cervical mobility through a wide range of therapeutic procedures, including mobilization or manipulation techniques. Previous systematic reviews reported preliminary evidence for the application of upper cervical manual therapy techniques for the management of headache.

The objective of this study is to study the effects of upper cervical translatoric spinal mobilization (UC-TSM) on headache intensity, cervical mobility and pressure pain threshold in subjects with headache. For this purpose, the investigators will conduct a randomized controlled trial. Volunteers with headache will participate in the study and will be randomly divided into control or treatment group. Treatment group will receive UC-TSM and the control group will receive no treatment.

Headache intensity, cervical mobility, temporomandibular mobility and pressure pain thresholds (PPT) will be measured before and immediately after each treatment session (3 treatment sessions in one week period) and after one month follow-up. At this moment, global perceived effect will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Present a history of headache.

Exclusion Criteria:

* Receive cervical treatment in the previous month.
* Present red flags for headache.
* Present any contraindications to manual therapy.
* Current involvement in compensations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Headache intensity as measured by Visual Analog Scale | From Baseline to one month follow-up

SECONDARY OUTCOMES:
Cervical mobility as measured by cervical range of motion device (CROM) | 1 minute Pre-Intervention, 1 minute Post-Intervention, One month follow-up
Pressure pain threshold as measured by digital algometer (Somedic Farsta) | 1 minute Pre-Intervention, 1 minute Post-Intervention, One month follow-up
Temporomandibular joint mobility as measured by digital calipher (mouth opening) | 1 minute Pre-Intervention, 1 minute Post-Intervention, One month follow-up
Global Perceived Effect as measured by Global Perceived Effect Scale (-5 to +5 Likert Scale) | One month follow-up
Immediate headache intensity changes as measured by Visual Analog Scale | 1 minute Pre-Intervention, 1 minute Post-Intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad de Investigación en Fisioterapia, Zaragoza, Aragon, Spain

REFERENCES:
- [Derived] Malo-Urries M, Tricas-Moreno JM, Estebanez-de-Miguel E, Hidalgo-Garcia C, Carrasco-Uribarren A, Cabanillas-Barea S. Immediate Effects of Upper Cervical Translatoric Mobilization on Cervical Mobility and Pressure Pain Threshold in Patients With Cervicogenic Headache: A Randomized Controlled Trial. J Manipulative Physiol Ther. 2017 Nov-Dec;40(9):649-658. doi: 10.1016/j.jmpt.2017.07.007. PMID 29229055